CLINICAL TRIAL: NCT02613598
Title: Phase I Dose Escalation Study to Determine the Maximum Tolerated Dose of the Combination of Ruxolitinib and Bortezomib in Patients With Relapsed or Refractory Lymphoma
Brief Title: Dose Escalation Study to Determine the Maximum Tolerated Dose of the Combination of Ruxolitinib and Bortezomib in Patients With Relapsed or Refractory Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2014.066; HUM00104716 (Other: University of Michgan Medical School)
Record Dates: First submitted 2015-11-20; First posted 2015-11-24 (Estimated); Last update posted 2021-12-20 (Actual); Status verified 2021-12

CONDITIONS: Hodgkin's Lymphoma; Lymphoma, Non-Hodgkin
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, Non-Hodgkin | interventions — Bortezomib; ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Bortezomib and Ruxolitinib (Experimental): Bortezomib on days 1, 4, 8, and 11 of a 21 day cycle in combination with Ruxolitinib (5, 10, 15, 20, or 25 mg) twice daily.
  Interventions: Drug: Bortezomib; Drug: Ruxolitinib

INTERVENTIONS:
Drug: Bortezomib
  Other Names: Velcade
Drug: Ruxolitinib
  Other Names: Jakafi

SUMMARY:
The primary objective of this research study is to determine the maximum tolerated dose (MTD) of Ruxolitinib (Jakafi) in combination with standard dose Bortezomib (Velcade) in patients with relapsed or refractory Hodgkin (HL) and Non-Hodgkin Lymphoma (NHL).

DETAILED DESCRIPTION:
Treatment of relapsed and refractory Hodgkin and Non-Hodgkin's Lymphoma remains difficult. To improve upon current efficacy rates new treatment modalities are needed. Currently modalities based upon targeting specific pathway and molecular receptors have made the greatest impact in the outcomes of refractory patients.

The JAK-Stat pathway and NF-κB are two such targets that have been shown to fuel the malignant transformation and growth of both myeloma and lymphoma. Blockade of key points in these molecular pathways has the potential of halting the pro-survival machinery. Combined inhibition of JAK/Stat and NF-κB may lead to synergistic effects as well as possibly mitigating some of the mechanisms of resistance to either agent. In this proposal, the investigators aim to utilize the JAK/Stat inhibitor ruxolitinib (Jakafi) and proteasome inhibitor bortezomib (Velcade) to target two major pathways of malignant transformation in hematologic malignancies.

The primary objective of this research study is to determine the maximum tolerated dose (MTD) of Ruxolitinib (Jakafi) in combination with standard dose Bortezomib (Velcade) in patients with relapsed or refractory Hodgkin (HL) and Non-Hodgkin Lymphoma (NHL).

The University of Michigan will enroll 24 subjects. Eligible subjects will have histologically or cytologically confirmed Hodgkin and Non-hodgkin's Lymphoma excluding Burkitt, CLL and lymphoblastic lymphoma that is considered to have relapsed or to be refractory to primary chemotherapy. Any prior exposure to Jakafi is excluded.

ELIGIBILITY:
Inclusion Criteria:

* Women and men with histologically or cytologically confirmed Hodgkin and all NHL subtypes excluding Burkitt, CLL and lymphoblastic lymphoma that is considered to have relapsed or to be refractory to primary chemotherapy.
* No previous anti-cancer therapy for at least 21 days and recovered from all treatment related toxicity
* Prior radiation is allowed prior to study start (1st dose of study medication) if at least 21 days have elapsed since prior large-field radiation therapy and all treatment related toxicity has resolved. At least 3 months must have passed since radio-immunotherapy.
* Prior auto graft is allowed prior to study start (1st dose of study medication), but patients must be at least 3 months from date of stem cell infusion and have recovered to ≤ grade 1 toxicities related to this procedure.
* Prior allogeneic transplants is allowed prior to study start (1st dose of study medication), but patients must be at least 6 months from date of stem cell infusion, have no evidence of GVHD, be off all immunosuppressant medications, and have recovered to ≤ grade 1 toxicities related to this procedure.
* Age >18 years
* ECOG (Eastern Cooperative Oncology Group) Performance status ≤2
* Life expectancy without treatment > 12 weeks
* Patients must have adequate hematologic, hepatic, and renal function as defined as: Absolute neutrophil count ≥1,000/μl, Platelets ≥75,000/μl, (50,000/ μl if due to BM involvement), Direct bilirubin< 1.5 mg/dl, unless due to Gilbert's or secondary to hemolysis, AST (Aspartate Aminotransferase) and/or ALT (Alanine Transaminase) <2.5 X institutional upper limit of normal unless due to lymphomatous involvement of the liver, Creatinine < 1.5 mg/dl and/or creatinine clearance >60 mL/min using the Cockcroft-Gault formula and no symptoms attributable to grade 2 or higher peripheral neuropathy.
* Should a woman become pregnant or suspect that she is pregnant while she or her partner is participating in this study, she should inform the treating physician immediately.
* Subjects must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients who are currently receiving any other experimental agent, patients must have stopped other experimental agents at least 21 days prior to 1st study dose.
* Any prior to exposure to Jakafi
* Patients with untreated brain metastases are excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to Jakafi or Velcade.
* Patients with uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant or breastfeeding women are excluded from this study because Jakafi is inhibitor of the Jak-1 and Jak-2 kinases with the potential for teratogenic or abortifacient effects. Because there is an unknown, but potential risk for adverse events in nursing infants secondary to treatment of the mother with Jakafi, breastfeeding should be discontinued if the mother is treated with Jakafi. These potential risks may also apply to other agents used in this study.
* HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with Jakafi. In addition, these patients are at increased risk of lethal infections when treated with marrow suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.
* Patients with grade 2 or higher peripheral neuropathy are excluded.
* Patients with CLL (Chronic Lymphocytic Leukemia), Burkitt or lymphoblastic lymphoma are excluded.
* Patients who would be required to concurrently take ruxolitinib in conjunction with a strong CYP3A4 inhibitors and have a platelet count less than 100,000 are ineligible for the study.
* Patient who are required to take a strong CYP3A4 inducer are excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-05-12 (Actual); Primary Completion 2021-06-07 (Actual); Study Completion 2021-06-07 (Actual)

PRIMARY OUTCOMES:
The Maximum Tolerated Dose (MTD) of Ruxolitinib in Combination with Standard Dose Bortezomib | Up to 5 Years

CONTACTS AND LOCATIONS:
Overall Officials: Tycel Phillips, M.D., Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michgan Comprehensive Cancer Center, Ann Arbor, Michigan, United States